CLINICAL TRIAL: NCT03823079
Title: A Randomized Phase II Study of Recombinant Human Thrombopoietin (Rh-TPO) and Recombinant Human Interleukin-11 (rhIL-11) for Recurrent Colorectal Cancer (CRC) Patients With Thrombocytopenia
Brief Title: Comparison of Interleukin-11 and rhTPO for Recurrent Colorectal Cancer Patients With Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-009
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Colorectal Carcinoma; Thrombopenia
Keywords: Recombinant human interleukin-11; Recombinant human thrombopoietin
MeSH Terms: conditions — Colorectal Neoplasms; Thrombocytopenia | interventions — Irinotecan; raltitrexed; Radiotherapy; oprelvekin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTPO arm (Experimental): rhTPO: 300 u/kg, subcutaneous injection, per day. (stopped as soon as the platelet count rises to normal)
  Concurrent Chemoradiotherapy:
  Radiation: judged according to the tumor site and radiotherapy purpose.
  Irinotecan: 80 mg/m2 (UGT1A1*28 6/6) or 65 mg/m2 (UGT1A1*28 6/7)
  Raltitrexed: 3 mg/m2 q3w
  Interventions: Drug: rhTPO; Drug: irinotecan; Drug: Raltitrexed; Radiation: radiotherapy
- rhIL-11 arm (Active Comparator): rhIL-11: 50 ug/kg, subcutaneous injection, per day. (stopped as soon as the platelet count rises to normal)
  Concurrent Chemoradiotherapy:
  Radiation: judged according to the tumor site and radiotherapy purpose.
  Irinotecan: 80 mg/m2 (UGT1A1*28 6/6) or 65 mg/m2 (UGT1A1*28 6/7)
  Raltitrexed: 3 mg/m2 q3w
  Interventions: Drug: irinotecan; Drug: Raltitrexed; Radiation: radiotherapy; Drug: rhIL-11

INTERVENTIONS:
Drug: rhTPO — rhTPO 300u/kg, subcutaneous injection, qd
  Arms: rhTPO arm
Drug: irinotecan — 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
Drug: Raltitrexed — 3mg/m2 q3w
Radiation: radiotherapy — in the use of intensity-modulated radiotherapy (IMRT) technology, the dose is judged according to the tumor site and radiotherapy purpose.
Drug: rhIL-11 — rhIL-11 50ug/kg, subcutaneous injection, qd
  Arms: rhIL-11 arm

SUMMARY:
This randomized controlled clinical phase II study was designed to compare the effect of rhTPO with rhIL-11 in improving thrombocytopenia in patients with recurrent colorectal cancer who underwent radiotherapy and with thrombocytopenia.

DETAILED DESCRIPTION:
Most patients with recurrent CRC have undergone a six-month postoperative adjuvant chemotherapy with oxaliplatin plus fluorouracil. Although the main dose-limiting side effect of oxaliplatin is neurotoxicity, with the widespread use of this drug, there are more and more reports that oxaliplatin is discontinued because of thrombocytopenia, which increases the risk of bleeding, rate of blood transfusion needs and length of stay. On the other hand, patients undergoing pelvic radiotherapy may also experience significant bone marrow suppression because flat bones such as the tibia may be exposed to high doses radiation. Low platelet counts is an urgent problem to be solved in order to give adequate quantitative radiotherapy. This randomized controlled clinical phase II study was designed to compare the effect of rhTPO with rhIL-11 in improving thrombocytopenia in patients with recurrent colorectal cancer who underwent radiotherapy and with thrombocytopenia, thus providing more evidence in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The primary tumor is colorectal cancer, histologically proved recurrence or metastasis disease, or pelvic relapse within 6 months after oxaliplatin-based adjuvant chemotherapy.
* Not suitable for re-use of oxaliplatin and fluorouracil.
* No medication history of irinotecan.
* Lesions evaluable, and has indications for radiotherapy.
* UGT1A1*28 gene phenotype is 6/6 or 6/7
* Karnofsky physical condition score ≥ 70
* Baseline platelet counts are 25-75×10^9/L, other bone marrow reserve and liver and kidney function meet the requirements of radiotherapy
* Able to follow the program during the study period
* Sign the informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Those with other history of malignant disease in the past 5 years, except for cured skin cancer and cervical carcinoma in situ
* If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
* Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months
* Organ transplantation requires immunosuppressive therapy
* Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
* Subject blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP) ≤2.5 times the normal upper limit; serum total bilirubin <1.5 times the normal upper limit; serum creatinine <1 times the normal upper limit; serum albumin ≥ 30g / L
* Anyone who is allergic to any research medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
the rate of recovery of platelet accounts | From date of chemoradiation until the date of first documented recovery, assessed up to 6 months
the duration after returning to normal | From date of first documented recovery until the date of first documented decrease of platelet accounts, assessed up to 6 months

SECONDARY OUTCOMES:
cycles of concurrent chemotherapy patients received during radiotherapy | through chemoradiation, an average of 5 weeks
change of participant quality of life during treatment as assessed by EORTC-quality of life questionnaire-C30 | at the beginning and the end of chemoradiation.
change of participant quality of life during treatment as assessed by EuroQol-5 dimensional (EQ-5D) questionnaire | at the beginning and the end of chemoradiation.
the rate of pathological complete response. | Surgery scheduled 6-8 weeks after the end of chemoradiation
  pathological complete response (pCR) was defined no viable cancer cell under the examination of surgical resection specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Study Chair — Fudan University

IPD SHARING:
Plan to Share IPD: No